CLINICAL TRIAL: NCT04062266
Title: Phase II Study of 5-Azacytidine (AZA) + Venetoclax as Maintenance Therapy in Patients With AML in Remission
Brief Title: AZA + Venetoclax as Maintenance Therapy in Patients With AML in Remission
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0226; NCI-2019-04987 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0226 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-08-16; First posted 2019-08-20 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia in Remission; FLT3 Gene Mutation; Hematologic and Lymphocytic Disorder; Acute Myeloid Leukemia; Minimal Residual Disease Persistence; Therapy-Related Acute Myeloid Leukemia
MeSH Terms: conditions — Hematologic Diseases; Leukemia, Myeloid, Acute | interventions — Azacitidine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (azacytidine, venetoclax) (Experimental): Patients receive azacitidine SC or IV over 1 hour daily on days 1-5, and venetoclax PO daily on days 1-14. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Given SC or IV
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial studies how well azacitidine and venetoclax work in treating patients with acute myeloid leukemia that is in remission. Drugs used in chemotherapy, such as azacitidine and venetoclax, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess relapse-free survival (RFS) of patients (pts) with acute myeloid leukemia (AML) treated with 5-azacytidine (azacitidine; AZA) combined with venetoclax (VEN) as maintenance therapy after achieving remission.

SECONDARY OBJECTIVES:

I. To assess modified RFS of pts with AML treated with 5-azacytidine combined with venetoclax as maintenance therapy.

II. To assess overall survival (OS) of pts with AML treated with 5-azacytidine combined with venetoclax as maintenance therapy.

III. To assess event-free survival (EFS) of pts with AML treated with 5-azacytidine combined with venetoclax as maintenance therapy.

IV. To assess the duration of remission (CRd) of pts with AML treated 5-azacytidine combined with venetoclax as maintenance therapy.

V. To assess toxicity and safety of 5-azacytidine combined with venetoclax as maintenance therapy in pts with AML.

VI. To assess the effects of 5-azacytidine combined with venetoclax on dynamics of minimal residual disease (MRD) and their relationship to outcomes.

OUTLINE:

Patients receive azacitidine subcutaneously (SC) or intravenously (IV) over 1 hour daily on days 1-5, and venetoclax orally (PO) daily on days 1-14. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 6-12 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged >/= 18 years AML who have achieved their FIRST CR or CRi and are not immediately candidates for allogeneic stem cell transplant.
2. Patients who have received intensive therapy (defined as receiving standard or higher dose cytarabine-based therapy) to achieve remission (CR/CRi) should have received remission induction therapy and at least 1 consolidation cycle. These patients are eligible as long as they are not greater than 2 months from their last consolidation therapy and will be enrolled in COHORT 1.
3. Patients who have received lower intensity therapy (defined as receiving low-dose cytarabine (LDAC) or hypomethylating agent (HMA)-based therapy) to achieve remission should have received at least 2 cycles of lower intensity therapy between the time they have achieved CR/CRi and enrollment on this protocol. They will be treated on COHORT 2.
4. For either subgroup (lower or higher intensity), patients who have measurable residual disease may be enrolled on their respective cohort at any time without maximum 'time from consolidation' requirement.
5. ECOG performance status of < or = 3
6. Adequate organ function as follows:

   1. Serum total bilirubin < or = to 1.5 X the Upper Limit of Normal (ULN)
   2. Serum creatinine < or = to 2.5 x ULN
7. Adequate BM reserve:

   1. Absolute neutrophil count (ANC) > 0.5 x k/uL
   2. Platelet count > or = 30 x k/uL
8. For females of childbearing age, they may participate if they:

   1. Have a negative serum or urine pregnancy test within 10 to 14 days of enrolling
   2. Agree to either abstinence or 2 effective contraceptive methods (such as barrier methods or hormonal contraception) throughout the treatment period and up to 30 days after discontinuing treatment.
9. For male patients with a female partner of childbearing age, they may participate if they agree to either abstinence or 2 effective contraceptive methods throughout the treatment period and up to 30 days after discontinuing treatment.
10. Ability to understand and sign informed consent.

Exclusion Criteria:

1. Diagnosis of acute promyelocytic leukemia (APL), AML - M3 by FAB classification based on morphology, immunophenotype, molecular, or cytogenetic s studies.
2. Diagnosis of AML associated t(15;17) or APL variant. Patients with t(9;22) are also ineligible unless they are unable or unwilling to receive therapy with a tyrosine kinase inhibitor.
3. Uncontrolled intercurrent illness including, but not limited to active uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
4. Patients with active CNS (central nervous system) disease.
5. Patients with documented hypersensitivity to any components of the study program.
6. Females who are pregnant or lactating or intending to become pregnant during the study.
7. Patients with history of extramedullary AML, except for CNS involvement that is currently controlled, will not be eligible for enrollment.
8. Patient should be removed from current trial if they wish to participate and get treatment on another trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-09-13 (Actual); Primary Completion 2030-10-31 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival (RFS) | From date of complete remission (CR) or complete remission with incomplete count recovery (CRi), assessed for up to 10 years
  The study will be continuously monitored for the primary endpoint, RFS, using the method of Thall, Wooten, and Tannir (2005). Will also summarize the posterior distribution of lambda-E (i.e., median RFS) assuming posterior mean and 95% credible interval.

SECONDARY OUTCOMES:
Incidence of toxicity | Up to 10 years
  Toxicities are defined as any treatment -related clinically significant grade 3 or 4 non-hematologic adverse events occurred during cycles 1-2 of the trial. Will continuously monitor treatment-related toxicities using the Bayesian approach of Thall, Simon, Estey (1995).
Modified RFS | Time from enrollment on study until date of first objective documentation of relapse or death, assessed for up to 10 years
  Distribution assessed using Kaplan-Meier method.
Overall survival (OS) | From the start of study treatment until date of death due to any cause, assessed for up to 10 years
  Distribution assessed using Kaplan-Meier method.
Event free survival (EFS) | From the start of study treatment until date of first confirmed relapse, withdrawal from study due to adverse event, or death due to any cause, assessed for up to 10 years
  Distribution assessed using Kaplan-Meier method.
Complete remission duration (CRd) | Time from CR or CRi until date of first objective documentation of confirmed relapse, assessed for up to 10 years
  Distribution assessed using Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Tapan M Kadia, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Bazinet A, Kantarjian H, Bataller A, Pemmaraju N, Borthakur G, Chien K, Alvarado Y, Bose P, Jabbour E, Yilmaz M, DiNardo C, Issa G, Montalban-Bravo G, Short N, Sasaki K, Bull-Linderman D, Daver N, Garcia-Manero G, Ravandi F, Kadia T. Reduced dose azacitidine plus venetoclax as maintenance therapy in acute myeloid leukaemia following intensive or low-intensity induction: a single-centre, single-arm, phase 2 trial. Lancet Haematol. 2024 Apr;11(4):e287-e298. doi: 10.1016/S2352-3026(24)00034-6. PMID 38548404
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org